CLINICAL TRIAL: NCT01760473
Title: Reinforcing Effects of Intranasal Buprenorphine Versus Buprenorphine/Naloxone in Buprenorphine-maintained Intranasal Drug Users
Brief Title: Reinforcing Effects of Intranasal (IN) Buprenorphine Versus Buprenorphine/Naloxone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #5879
Record Dates: First submitted 2009-05-01; First posted 2013-01-04 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Heroin Dependence
Keywords: opioid dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: In this study's design, all participants received each of the 9 intranasal test drugs under investigation. This study employed a Latin-square randomization procedure, therefore, the sequence of testing for the 9 intranasal drugs was unique for each participant.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Bup 8 (Experimental): Intranasal challenge drug: 8 mg of Buprenorphine administered intranasally.
  Interventions: Drug: Intranasal challenge drug
- Bup 16 (Experimental): Intranasal challenge drug: 16 mg of Buprenorphine administered intranasally.
  Interventions: Drug: Intranasal challenge drug
- Bup/Nal 8/2 (Experimental): Intranasal challenge drug: 8 mg of Buprenorphine administered intranasally with 2 mg of Naloxone.
  Interventions: Drug: Intranasal challenge drug
- Bup/Nal 8/8 (Experimental): Intranasal challenge drug: 8 mg of Buprenorphine administered intranasally with 8 mg of Naloxone.
  Interventions: Drug: Intranasal challenge drug
- Bup/Nal 8/16 (Experimental): Intranasal challenge drug: 8 mg of Buprenorphine administered intranasally with 16 mg of Naloxone.
  Interventions: Drug: Intranasal challenge drug
- Bup/Nal 16/4 (Experimental): Intranasal challenge drug: 16 mg of Buprenorphine administered intranasally with 4 mg of Naloxone.
  Interventions: Drug: Intranasal challenge drug
- Heroin (Active Comparator): Intranasal challenge drug: 24 mg of heroin administered intranasally.
  Interventions: Drug: Intranasal challenge drug
- Placebo (Sham Comparator): Intranasal challenge drug: Intranasal lactose powder.
  Interventions: Drug: Intranasal challenge drug
- Naloxone 4 mg (Active Comparator): Intranasal challenge drug: Intranasal Naloxone 4mg.
  Interventions: Drug: Intranasal challenge drug

INTERVENTIONS:
Drug: Intranasal challenge drug — Each of the experimental challenge drugs were administered intranasally to all participants in random order.

SUMMARY:
The study is designed to compare the abuse liabilities of intranasal buprenorphine and buprenorphine/naloxone in individuals who are physically dependent on sublingual buprenorphine. The investigators hypothesize that the abuse liability of buprenorphine/naloxone is lower than that of buprenorphine alone.

DETAILED DESCRIPTION:
Although sublingual buprenorphine is an effective treatment for opioid addiction, the medication itself has abuse liability and, in some countries, has largely replaced heroin as the opioid drug of choice. In response to the reports of diversion and abuse of sublingual (SL) buprenorphine, a potentially less abusable formulation of buprenorphine that contains naloxone is being marketed in several countries. However, the relative abuse liability of buprenorphine alone and the buprenorphine/naloxone combination in buprenorphine-dependent individuals is unclear. Preliminary data from a study funded by Schering-Plough Corporation suggest that the buprenorphine/naloxone combination, when given intravenously (IV), does indeed have less abuse liability than IV buprenorphine in buprenorphine-dependent individuals. In addition to IV abuse of buprenorphine, epidemiological data suggest that buprenorphine is widely abused by the intranasal (IN) route. However, no data exist on the abuse liability of either IN buprenorphine alone or the buprenorphine/naloxone combination. Several studies have shown that naloxone is an effective antagonist of opioid agonist effects when given intravenously, but it is not clear whether naloxone given intranasally is as effective as when it is given by other routes of administration. Some studies have suggested that they are equally effective (Loimer et al., 1994), but others have shown that naloxone given intranasally is less effective (i.e., has a slower onset of effects) than when given by other routes of administration (Kelly et al., 2005). How this may impact on the ability of naloxone to reduce the reinforcing effects of IN buprenorphine is unclear. The primary aim of the current study proposal is to compare the reinforcing effects of IN buprenorphine and buprenorphine/naloxone in IN opioid abusers who are maintained on SL buprenorphine using a study design parallel to that used in our recent studies of the abuse liability of IV buprenorphine and buprenorphine/naloxone. Placebo, heroin, and naloxone will be used as neutral, positive, and negative controls, respectively. Secondary aims are to compare the subjective, performance, and physiological effects of IN buprenorphine and buprenorphine/naloxone. Overall, this study will complement our investigations of IV buprenorphine products by allowing for a complete overview within the same laboratory self-administration model of both the intravenous and intranasal abuse liability of buprenorphine versus buprenorphine/naloxone in individuals maintained on buprenorphine. The primary aim of the study is to compare the reinforcing effects of IN buprenorphine and IN buprenorphine/naloxone in opioid abusers maintained on different doses of sublingual buprenorphine. Secondary aims of the study are to compare the subjective, performance and physiological effects of IN buprenorphine and IN buprenorphine/naloxone. IN-administered placebo (lactose powder), naloxone alone, and heroin alone will be tested as neutral, negative, and positive control conditions, respectively. Participants (N=12 completers) will reside on an inpatient unit (5-South) during a 7 to 8-week study. This research will provide useful information to clinicians treating opioid dependent individuals with buprenorphine, and importantly, will provide information about the abuse potential and effects of buprenorphine on multiple measures of human functioning.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV criteria for heroin dependence
* No major mood, psychotic, or anxiety disorder
* Physically healthy
* Able to perform study procedures
* 21-45 years of age
* Normal body weight
* Current use of opioids in amounts and/or frequencies that meet or exceed those used in the proposed study (e.g., 1-2 bags of heroin per occasion at least twice per day)
* Self-administer IN buprenorphine above placebo levels during the qualification phase (see below)

Exclusion Criteria:

* DSM IV criteria for dependence on drugs other than opioids, nicotine or caffeine
* Participants requesting treatment
* Participants on parole or probation
* Pregnancy or lactation
* Birth, miscarriage or abortion within 6 months
* Current or recent history of significant violent behavior
* Current major Axis I psychopathology, other than opioid dependence (e.g., mood disorder with functional impairment or suicide risk, schizophrenia), that might interfere with ability to participate in the study
* AST or ALT > 3 times the upper limit of normal
* Significant suicide risk
* Current chronic pain
* Sensitivity, allergy, or contraindication to opioids
* Current or recent (past 30 days) physical dependence on or treatment with methadone, buprenorphine, or the buprenorphine/naloxone combination

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Comer, PHD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute and Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Challege Drug: Each of the 9 experimental challenge drugs were administered intranasally to all participants in random order. This study employed a Latin-square randomization procedure, therefore, the testing order of the 9 IN doses was unique for each participant.
Period: Overall Study
Arm/Group | Intranasal Challege Drug
Started | 27
Completed | 12
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Intranasal Challege Drug: Each of the 9 experimental challenge drugs were administered intranasally to all participants in random order.
Arm/Group | Intranasal Challege Drug
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Drug Self-administration
Description: The maximum number of responses (clicks on a computer mouse) the participant was willing to perform in order to receive a dose of the intranasal challenge drug under investigation.
Time Frame: Throughout the testing sessions (approximately 9 weeks).
Measure: Mean (Standard Error); unit: Clicks on a computer mouse
Arm/Group | Bup 8 | Bup 16 | Bup/Nal 8/2 | Bup/Nal 8/8 | Bup/Nal 8/16 | Bup/Nal 16/4 | Heroin | Placebo | Naloxone 4 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Clicks on a computer mouse | 350 (135) | 255 (121) | 223 (113) | 113 (83) | 2.7 (2.7) | 191 (112) | 755 (156) | 38 (23) | 45 (30)

2. Secondary Outcome: SOWS
Description: Subjective opioid withdrawal scale (SOWS) measure (0-64). Greater score indicates more severe withdrawal.
Time Frame: Throughout the testing sessions (approximately 9 weeks).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bup 8 | Bup 16 | Bup/Nal 8/2 | Bup/Nal 8/8 | Bup/Nal 8/16 | Bup/Nal 16/4 | Heroin | Placebo | Naloxone 4 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
units on a scale | 3 (.5) | 3 (.7) | 3 (.9) | 3 (.8) | 5 (1) | 3 (.5) | 2 (.3) | 2 (.53) | 7 (1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day of admission until discharge and at 3 month follow-up
Groups:
- Intranasal Challege Drug: Each of the 9 experimental challenge drugs were administered intranasally to all participants in a randomized order. Therefore, the testing sequence for each of the participants was unique. Although we assessed for some averse events on a daily basis, other measures of health (e.g., blood chemistry) were assessed on a weekly basis. As multiple doses were tested during the week, therefore, in some cases we cannot causally connect some AEs to any individual drug/testing condition.
Arm/Group | Intranasal Challege Drug
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Challege Drug (N=27)
Elevated liver function test (AST/ALT) (Metabolism and nutrition disorders) | 2 (2) — Liver function rose to greater than 3 x the upper limit of normal. Blood chemistry was performed on a weekly basis throughout the 9 weeks. As multiple doses were tested during the week, we cannot attribute this AE to any individual drug condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No